CLINICAL TRIAL: NCT03696251
Title: The Current Situation and Prospects of Master's Nursing Programs in Taiwan
Brief Title: Master's Nursing Programs in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201807093RINB
Record Dates: First submitted 2018-09-30; First posted 2018-10-04 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-09

CONDITIONS: Master's Nursing Programs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- master's nursing program: the graduates of master's nursing program in recent three years in Taiwan

SUMMARY:
The purpose of the study: (1) to understand the models of master education in nursing in Taiwan, including goals, curriculum, and clinical hours…etc). (2) to explore the clinical competencies and career development of the graduates of master's nursing program in Taiwan. Methods: Researchers will collect the data of program goals, curriculum, and clinical hours…etc. from the websites of all nursing schools that provide master's education in nursing in Taiwan. A structured self-report questionnaire will be used to collect the data of the clinical competence and career development of the graduates who have graduated from a master's nursing program in Taiwan in recent 3 years. A third of all eligible subjects will be randomly selected and invited to fill out the questionnaire by the schools that they graduated from.

ELIGIBILITY:
Inclusion Criteria:

1. the graduates who have graduated from a master's nursing program in Taiwan in recent 3 years (2015-2017)
2. The persons who are willing to participate in the study and fill out the questionnaire.

Exclusion Criteria:

1. The person who is unable to read and write Chinese.
2. The person who is unable to fill out the questionnaire by him/her-self

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: the graduates who have graduated from a master's nursing program in Taiwan in recent 3 years.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2018-12-15 (Estimated); Study Completion 2018-12-15 (Estimated)

PRIMARY OUTCOMES:
clinical competencies of study subjects | up to 24 weeks
  Clinical Nurse Specialist Core Competencies Questionnaire will be used for measuring clinical competencies of study subjects. There are 67 items in the questionnaire. The questionnaire employ 5 point Likert-scale. The subject will be asked to assess his/her own clinical competence and choose an appropriate number for each item. The higher number means higher level of clinical competence.

SECONDARY OUTCOMES:
The questionnaire of employment status | up to 24 weeks
  Study subjects will be asked to fill out whether they are active practice nurse and the information of their current job, including workplace (such as hospital, community health center, school,…etc.), current job title (such as staff nurse, head nurse, nurse supervisor, clinical instructor, nurse practitioner,…etc.) and full-time or part-time.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided